CLINICAL TRIAL: NCT02182947
Title: Comparison of the Use of Wireless Capsule Endoscopy With Magnetic Resonance Enterography in Children With Inflammatory Bowel Disease
Brief Title: Capsule Endoscopy in Inflammatory Bowel Disease (IBD) in Children
Acronym: CE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Mercy Hospital Kansas City (Other)
Collaborators: Medtronic - MITG (Industry)
Responsible Party: Principal Investigator, Nadia Hijaz, MD, Children's Mercy Hospital Kansas City
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 13080263
Record Dates: First submitted 2014-06-30; First posted 2014-07-08 (Estimated); Results first posted 2021-03-11 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2021-02

CONDITIONS: IBD
Keywords: Pediatric; Inflammatory Bowel Disease; Wireless capsule endoscopy; MRE; Crohn's Disease; Indeterminant Colitis; Small bowel Crohn's Disease
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease | interventions — Capsule Endoscopy; Endoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Endoscopy Imaging (Experimental): Wireless-video capsule endoscopy (WCE) compared to the findings of MRE magnetic resonance enterography in same group of patients.
  Interventions: Device: Capsule endoscopy

INTERVENTIONS:
Device: Capsule endoscopy — Pediatric patients with indeterminate colitis (IC) or Crohn's disease (CD) who are scheduled to undergo routine small bowel screening or surveillance using MRE. Subjects will swallow a patency capsule (PC) to study bowel patency.Those patients, who pass an intact PC, usually within 40 hours, will ingest the wireless capsule endoscopy (WCE). The WCE will be performed within 1 week of completion of MRE.
  Other Names: Wireless capsule endoscopy, Pillcam from given imaging

SUMMARY:
Most of the studies evaluating the roles of MRE and WCE conducted in pediatric patients have been retrospective with the main goal of making a diagnosis in patients with suspected IBD. The current study is the first prospective study in children with known IBD assessing the roles of MRE and WCE in identifying disease exacerbation. This study will help to identify if capsule endoscopy is superior or complementary to MRE in the evaluation of suspected disease exacerbation in IBD patients.

DETAILED DESCRIPTION:
Proximal small bowel (SB) involvement in CD is associated with a more aggressive disease course and an increased need for surgery.Therefore, accurate determination of SB involvement in pediatric CD is crucial for optimal patient management. Current clinical guidelines include suggested modalities to identify SB involvement and determine management plans. Available options include small bowel series, computed tomography enterography (CTE), small bowel wireless capsule endoscopy (WCE), gadolinium enhanced MRI imaging (GAD MRI), and small bowel contrast enhanced ultrasound (US). The choice of modality is largely determined by available resources, radiation exposure risk, and physician and institutional preferences. MRE and contrast enhanced US are radiation free, while other radiologic modalities entail a risk of radiation exposure. WCE may entail a risk of capsule retention. The risk of capsule retention resulting in obstruction is increased in the context of stricturing or fistulizing disease in CD and has been estimated at 2.6% but may be greatly mitigated by patency capsule screening.

Magnetic resonance enterography (MRE) and small bowel contrast ultrasound (SICUS) have diagnostic effectiveness comparable to other radiological modalities for evaluation of CD patients. However, both studies have their own limitations, MRE is limited by expense, the availability of the requisite equipment and software, variable expertise in interpretation of the findings, and (potentially) the need for sedation in pediatric population. SICUS is similarly affected by being operator dependent with the requisite need of accumulated expertise and heightened need for cooperation during the study that can limit its use in pediatric populations.

Several diagnostic modalities have been evaluated in comparison to WCE in several pediatric and adult IBD studies. The studies conducted in children with IBD were mostly retrospective and aimed at evaluating the role of MRE and WCE for detection of SB disease. They concluded that MRE and WCE were comparable with similar sensitivities. Only three prospective studies (all European) in pediatric IBD have compared WCE and MRE modalities in identifying SB disease involvement. Two were studies in established CD and one in suspected CD and again, they suggested that the tests appear complementary for detection of active CD. The current study is the a another prospective study in children with established IBD in the United States assessing the roles of MRE and WCE in identifying SB disease involvement in IBD. This study provides evidence for capsule endoscopy in the evaluation of established disease exacerbation in patients with IBD in relation to MRE.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 4 to 17.99 years at time of investigation
* IBD/CD and IBD/IC diagnosed based on standard clinical - histologic criteria
* Patient is scheduled to have MRE as standard of care for evaluation of disease severity/ complication.
* Signed permission/assent/consent

Exclusion Criteria:

* IBD diagnosis not established
* Recent intestinal tract surgery / resection involving small bowel
* Use of NSAIDs 4 weeks prior to the Capsule endoscopy study.
* Patients are on prokinetic medication.
* Swallowing disorders, esophageal stricture or patients unable to swallow the capsule.
* Presence of gastrointestinal obstruction or ileus.
* Patient with implanted electro-medical device or pacemakers.

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2012-08 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2018-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nadia M Hijaz, MD, Principal Investigator — Children's Mercy
Locations (1):
- Children Mercy Hospital and Clinics, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cuffari C, Dubinsky M, Darbari A, Sena L, Baldassano R. Crohn's jejunoileitis: the pediatrician's perspective on diagnosis and management. Inflamm Bowel Dis. 2005 Jul;11(7):696-704. doi: 10.1097/01.mib.0000166933.74477.69. PMID 15973125
- [Background] North American Society for Pediatric Gastroenterology, Hepatology, and Nutrition; Colitis Foundation of America; Bousvaros A, Antonioli DA, Colletti RB, Dubinsky MC, Glickman JN, Gold BD, Griffiths AM, Jevon GP, Higuchi LM, Hyams JS, Kirschner BS, Kugathasan S, Baldassano RN, Russo PA. Differentiating ulcerative colitis from Crohn disease in children and young adults: report of a working group of the North American Society for Pediatric Gastroenterology, Hepatology, and Nutrition and the Crohn's and Colitis Foundation of America. J Pediatr Gastroenterol Nutr. 2007 May;44(5):653-74. doi: 10.1097/MPG.0b013e31805563f3. PMID 17460505
- [Background] Levi Z, Fraser E, Krongrad R, Hazazi R, benjaminov O, meyerovitch J, Tal OB, Choen A, Niv Y, Fraser G. Factors associated with radiation exposure in patients with inflammatory bowel disease. Aliment Pharmacol Ther. 2009 Dec 1;30(11-12):1128-36. doi: 10.1111/j.1365-2036.2009.04140.x. PMID 19899197
- [Background] Deviere J, Hochberger J, Neuhaus H, Ponchon T, Eugenidis N, Neumann C, Ladas S. Recommendations of the ESGE workshop on Ethical, Clinical, and Economic Dilemmas Arising from the Implementation of New Techniques. First European Symposium on Ethics in Gastroenterology and Digestive Endoscopy, Kos, Greece, June 2003. Endoscopy. 2003 Sep;35(9):768-71. doi: 10.1055/s-2003-41587. No abstract available. PMID 12929027
- [Background] Jensen MD, Nathan T, Rafaelsen SR, Kjeldsen J. Diagnostic accuracy of capsule endoscopy for small bowel Crohn's disease is superior to that of MR enterography or CT enterography. Clin Gastroenterol Hepatol. 2011 Feb;9(2):124-9. doi: 10.1016/j.cgh.2010.10.019. Epub 2010 Nov 5. PMID 21056692
- [Background] Moy L, Levine J. Capsule endoscopy in the evaluation of patients with unexplained growth failure. J Pediatr Gastroenterol Nutr. 2009 May;48(5):647-50. doi: 10.1097/MPG.0b013e31818b0ac7. PMID 19367183
- [Background] Casciani E, Masselli G, Di Nardo G, Polettini E, Bertini L, Oliva S, Floriani I, Cucchiara S, Gualdi G. MR enterography versus capsule endoscopy in paediatric patients with suspected Crohn's disease. Eur Radiol. 2011 Apr;21(4):823-31. doi: 10.1007/s00330-010-1976-3. Epub 2010 Oct 5. PMID 20922391
- [Background] Di Nardo G, Oliva S, Ferrari F, Riccioni ME, Staiano A, Lombardi G, Costamagna G, Cucchiara S, Stronati L. Usefulness of wireless capsule endoscopy in paediatric inflammatory bowel disease. Dig Liver Dis. 2011 Mar;43(3):220-4. doi: 10.1016/j.dld.2010.10.004. Epub 2010 Nov 18. PMID 21093392
- [Background] Liao Z, Gao R, Xu C, Li ZS. Indications and detection, completion, and retention rates of small-bowel capsule endoscopy: a systematic review. Gastrointest Endosc. 2010 Feb;71(2):280-6. doi: 10.1016/j.gie.2009.09.031. PMID 20152309
- [Background] Herrerias JM, Leighton JA, Costamagna G, Infantolino A, Eliakim R, Fischer D, Rubin DT, Manten HD, Scapa E, Morgan DR, Bergwerk AJ, Koslowsky B, Adler SN. Agile patency system eliminates risk of capsule retention in patients with known intestinal strictures who undergo capsule endoscopy. Gastrointest Endosc. 2008 May;67(6):902-9. doi: 10.1016/j.gie.2007.10.063. Epub 2008 Mar 19. PMID 18355824
- [Background] Flamant M, Trang C, Maillard O, Sacher-Huvelin S, Le Rhun M, Galmiche JP, Bourreille A. The prevalence and outcome of jejunal lesions visualized by small bowel capsule endoscopy in Crohn's disease. Inflamm Bowel Dis. 2013 Jun;19(7):1390-6. doi: 10.1097/MIB.0b013e31828133c1. PMID 23552764
- [Background] Kopylov U, Nemeth A, Koulaouzidis A, Makins R, Wild G, Afif W, Bitton A, Johansson GW, Bessissow T, Eliakim R, Toth E, Seidman EG. Small bowel capsule endoscopy in the management of established Crohn's disease: clinical impact, safety, and correlation with inflammatory biomarkers. Inflamm Bowel Dis. 2015 Jan;21(1):93-100. doi: 10.1097/MIB.0000000000000255. PMID 25517597
- [Background] Ladas SD, Triantafyllou K, Spada C, Riccioni ME, Rey JF, Niv Y, Delvaux M, de Franchis R, Costamagna G; ESGE Clinical Guidelines Committee. European Society of Gastrointestinal Endoscopy (ESGE): recommendations (2009) on clinical use of video capsule endoscopy to investigate small-bowel, esophageal and colonic diseases. Endoscopy. 2010 Mar;42(3):220-7. doi: 10.1055/s-0029-1243968. Epub 2010 Mar 1. PMID 20195992
- [Background] Aloi M, Di Nardo G, Romano G, Casciani E, Civitelli F, Oliva S, Viola F, Maccioni F, Gualdi G, Cucchiara S. Magnetic resonance enterography, small-intestine contrast US, and capsule endoscopy to evaluate the small bowel in pediatric Crohn's disease: a prospective, blinded, comparison study. Gastrointest Endosc. 2015 Feb;81(2):420-7. doi: 10.1016/j.gie.2014.07.009. Epub 2014 Aug 10. PMID 25115363
- [Background] Pallotta N, Tomei E, Viscido A, Calabrese E, Marcheggiano A, Caprilli R, Corazziari E. Small intestine contrast ultrasonography: an alternative to radiology in the assessment of small bowel disease. Inflamm Bowel Dis. 2005 Feb;11(2):146-53. doi: 10.1097/00054725-200502000-00008. PMID 15677908
- [Background] Kovanlikaya A, Watson E, Hayward J, Beneck D, Sockolow R, Solomon A, Christos P, Brill PW. Magnetic resonance enterography and wireless capsule endoscopy in the evaluation of patients with inflammatory bowel disease. Clin Imaging. 2013 Jan-Feb;37(1):77-82. doi: 10.1016/j.clinimag.2012.03.011. Epub 2012 Jun 8. PMID 23206611
- [Background] Oliva S, Cucchiara S, Civitelli F, Casciani E, Di Nardo G, Hassan C, Papoff P, Cohen SA. Colon capsule endoscopy compared with other modalities in the evaluation of pediatric Crohn's disease of the small bowel and colon. Gastrointest Endosc. 2016 May;83(5):975-83. doi: 10.1016/j.gie.2015.08.070. Epub 2015 Sep 9. PMID 26363334
- [Background] Kopylov U, Yung DE, Engel T, Vijayan S, Har-Noy O, Katz L, Oliva S, Avni T, Battat R, Eliakim R, Ben-Horin S, Koulaouzidis A. Diagnostic yield of capsule endoscopy versus magnetic resonance enterography and small bowel contrast ultrasound in the evaluation of small bowel Crohn's disease: Systematic review and meta-analysis. Dig Liver Dis. 2017 Aug;49(8):854-863. doi: 10.1016/j.dld.2017.04.013. Epub 2017 Apr 27. PMID 28512034
- [Background] Bryant RV, Winer S, Travis SP, Riddell RH. Systematic review: histological remission in inflammatory bowel disease. Is 'complete' remission the new treatment paradigm? An IOIBD initiative. J Crohns Colitis. 2014 Dec;8(12):1582-97. doi: 10.1016/j.crohns.2014.08.011. Epub 2014 Sep 27. PMID 25267173
- [Background] Giles E, Barclay AR, Chippington S, Wilson DC. Systematic review: MRI enterography for assessment of small bowel involvement in paediatric Crohn's disease. Aliment Pharmacol Ther. 2013 Jun;37(12):1121-31. doi: 10.1111/apt.12323. Epub 2013 May 3. PMID 23638954

RESULTS

PARTICIPANT FLOW:
Groups:
- Overall Study: Pediatric patients with indeterminate colitis (IC) or Crohn's disease (CD) who are scheduled to undergo routine small bowel screening or surveillance using Magnetic Resonance Enterography (MRE). Subjects will swallow a patency capsule (PC) to study bowel patency.Those patients, who pass an intact Patency Capsule (PC), usually within 40 hours, will ingest the wireless capsule endoscopy (WCE). The WCE will be performed within 1 week of completion of MRE.Wireless-video capsule endoscopy (WCE) compared to the findings of MRE magnetic resonance enterography in same group of patients.
Period: Overall Study
Arm/Group | Overall Study
Started | 45
Completed | 27
Not Completed | 18
Not completed — Withdrawal by Subject | 7
Not completed — Lost to Follow-up | 3
Not completed — Failed screening activities | 8

BASELINE CHARACTERISTICS:
Arm/Group | Overall Study
Number analyzed (Participants) | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.46 (2.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 20
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race Unrecorded | 27
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 27
Body Mass Index BMI percentile of each IBD patients [Mean (Standard Deviation); unit: Percentile] — Percentile of each patient's Body Mass Index BMI which is recorded at the time of enrolling in the study.
  Percentile | 57 (32.9)
Pediatric Crohns Disease Activity Index PCDAI [Mean (Standard Deviation); unit: units on a scale] — PCDAI is a score of CD disease activity Lowest is zero indicate lowest disease activity Highest is 100 indicate highest disease activity
  units on a scale | 10.2 (12.5)
Duration of disease year [Mean (Standard Deviation); unit: years] | 1.7 (2.32)
Percentage of patients with biologics use with or without immune modulators [Number; unit: Percent of patients] | 44.4
Percentage of patients with inflammatory phenotype of IBD [Number; unit: Percent of patients] | 93
Percentage of patients with stricturing phenotype of IBD [Number; unit: Percent of patients] | 7

OUTCOME MEASURES:

1. Primary Outcome: Diagnostic Yield of Magnetic Resonance Enterography (MRE)
Description: The reported positive Magnetic Resonance Enterography (MRE) studies percentage in pediatric patients with known Inflammatory Bowel Disease (IBD) including Crohn's disease (CD) or indeterminate colitis (IC).
  Diagnostic yield DY of MRE that is the ability of a test to show positive findings to diagnose small bowel Crohns disease based on specified criteria used in the study.The study is positive if it has score of >3 of radiological findings of (SB wall thickness, SB wall enhancement , mucosal and serosal enhancement suggestive of mesenteric fatty infiltration, strictures, comb sign which is increased mesenteric vascularity adjacent to the inflamed bowel loop, reactive mesenteric lymphadenopathy, the presence of fistula, stricture or abscess and the number of SB segments involved).
Time Frame: 1.5 years
Population: The Diagnostic yield of of MRE were calculated based on how many positive MRE test( with score >3) divided by total number of MRE studies analyzed.
Measure: Number; unit: % Percentage of Diagnostic yeild
Arm/Group | Overall Study
Number analyzed (Participants) | 27
% Percentage of Diagnostic yeild | 52

2. Primary Outcome: Diagnostic Yield of Wireless Capsule Endoscopy (WCE)
Description: The reported positive Wireless Capsule Endoscopy (WCE) percentage in pediatric patients with known Inflammatory Bowel Disease (IBD) including Crohn's disease (CD) or indeterminate colitis (IC).
  Diagnostic yield of wireless capsule endoscopy is the ability of this test to detect abnormalities and diagnose positive small bowel crohns disease. The positive (or active) WCE is defined if clear abnormalities of the SB mucosa (ulcerations >3, erosions, polyps, vascular lesions, and bleeding lesions). White lesions within a crater with surrounding erythema were considered ulcers, whereas small superficial white lesions, even with surrounding erythema, were considered erosions.
Time Frame: 1.5 years
Population: The diagnostic yield of WCE were calculated based on how many positive SB capsule study detecting SB changes (as defined by positive WCE test) divided by total number of WCE studies analyzed.
Measure: Number; unit: % Percentage of Diagnostic yeild
Arm/Group | Overall Study
Number analyzed (Participants) | 27
% Percentage of Diagnostic yeild | 37

3. Secondary Outcome: Sensitivity of Magnetic Resonance Enterography (MRE)
Description: The sensitivity MRE in identifying patients with active vs. inactive CD and IC as defined by the Pediatric Crohn's disease activity index (PCDAI).
Time Frame: 1.5 years
Measure: Mean (95% Confidence Interval); unit: Percent sensitivity
Arm/Group | Overall Study
Number analyzed (Participants) | 27
Percent sensitivity | 100 [54.07 to 100]

4. Secondary Outcome: Sensitivity of Wireless Capsule Endoscopy (WCE)
Description: The sensitivity of WCE in identifying patients with active vs. inactive CD and IC as defined by the Pediatric Crohn's disease activity index (PCDAI)
Time Frame: 1.5 years
Measure: Mean (95% Confidence Interval); unit: Percent sensitivity
Arm/Group | Overall Study
Number analyzed (Participants) | 27
Percent sensitivity | 83.3 [35.88 to 99.58]

5. Secondary Outcome: Specificity of Magnetic Resonance Enterography (MRE)
Description: The specificity of MRE in identifying patients with active vs. inactive CD and IC as defined by the Pediatric Crohn's disease activity index PCDAI
Time Frame: 1.5 years
Measure: Mean (95% Confidence Interval); unit: Percent specificity
Arm/Group | Overall Study
Number analyzed (Participants) | 27
Percent specificity | 57.14 [28.86 to 82.34]

6. Secondary Outcome: Specificity of Wireless Capsule Endoscopy
Description: The specificity of WCE in identifying patients with active vs. inactive CD and IC as defined by the Pediatric Crohn's disease activity index PCDAI
Time Frame: 1.5 years
Measure: Mean (95% Confidence Interval); unit: Percent specificity
Arm/Group | Overall Study
Number analyzed (Participants) | 27
Percent specificity | 83.3 [35.88 to 99.58]

7. Secondary Outcome: Accuracy of Magnetic Resonance Enterography (MRE)Accuracy
Description: The accuracy of Magnetic Resonance Enterography (MRE) in pediatric patients with known Inflammatory Bowel Disease (IBD) including Crohn's disease (CD) or indeterminate colitis (IC) in reference to pediatric Crohn's disease activity index PCDAI.
Time Frame: 1.5 years
Measure: Mean (95% Confidence Interval); unit: Percent accuracy
Arm/Group | Overall Study
Number analyzed (Participants) | 27
Percent accuracy | 70 [45.72 to 88.11]

8. Secondary Outcome: Accuracy of Wireless Capsule Endoscopy (WCE)
Description: The accuracy of WCE in pediatric patients with known Inflammatory Bowel Disease (IBD) including Crohn's disease (CD) or indeterminate colitis (IC) in reference to pediatric Crohn's disease activity index PCDAI.
Time Frame: 1.5 years
Measure: Mean (95% Confidence Interval); unit: Percent accuracy
Arm/Group | Overall Study
Number analyzed (Participants) | 27
Percent accuracy | 80 [56.34 to 94.27]

ADVERSE EVENTS:
Time Frame: 1.5 years
Groups:
- Overall Study: Pediatric patients with indeterminate colitis (IC) or Crohn's disease (CD) who are scheduled to undergo routine small bowel screening or surveillance using Magnetic Resonance Enterography (MRE).
Arm/Group | Overall Study
All-Cause Mortality (participants affected / at risk) | 0/45
Serious Adverse Events (participants affected / at risk) | 0/45
Other Adverse Events (participants affected / at risk) | 0/45

LIMITATIONS AND CAVEATS:
Small patient population limits the ability to largely generalize these results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-31): https://cdn.clinicaltrials.gov/large-docs/47/NCT02182947/Prot_SAP_000.pdf